CLINICAL TRIAL: NCT05302817
Title: Functional Lung Avoidance Radiation Therapy Using Hyperpolarized Xenon-129 MRI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Regulatory compliance.
Sponsor: Xemed LLC (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 849026
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: lung cancer; non-small-cell lung cancer; radiation therapy; guided radiation therapy; functional lung avoidance; hyperpolarized xenon; HXe MRI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1: open trial for establishing safety and methodology. Phase 1, Part 1: 10 subjects enrolled for establishing methodology for guiding radiation therapy using HXe MRI. Radiation treatment will follow standard-of-care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard-of-care Radiation Therapy for lung cancer using HXe MRI for diagnosis. (Experimental): Patients with non-small cell lung cancer scheduled for radiation therapy will be voluntarily enrolled in this study, where they will have their lung ventilation and function imaged with hyperpolarized xenon MRI. The 3D HXe images will be used in determining a functional lung avoidance treatment map. However, for this part of the study, subjects will still follow the standard-of-care radiation treatment plan. At 6-month follow up the subjects will be imaged again with HXe to assess lung ventilation and function post-RT compared to baseline (pre-RT). Additionally, standard-of-care lung testing (DLCO, PFT) and quality-of-life questionnaires will be assessed at several time points during the study.
  Interventions: Combination Product: Hyperpolarized xenon MRI
- Guided Radiation Therapy for lung cancer using HXe MRI for functional lung avoidance and diagnosis. (Experimental): Patients with non-small cell lung cancer scheduled for radiation therapy will be voluntarily enrolled in this study. They will have their lung ventilation and function imaged with hyperpolarized xenon MRI. The 3D HXe images will be used in determining a functional lung avoidance treatment map. Patients will follow radiation therapy optimized for functional lung avoidance. At 6-month follow up the subjects will be imaged again with HXe to assess lung ventilation and function post-RT compared to baseline (pre-RT). Additionally, standard-of-care lung testing (DLCO, PFT) and quality-of-life questionnaires will be assessed at several time points during the study.
  Interventions: Combination Product: Hyperpolarized xenon MRI

INTERVENTIONS:
Combination Product: Hyperpolarized xenon MRI — Patients with non-small cell lung cancer scheduled for radiation therapy willing to take part in this study will undergo hyperpolarized xenon MRI at several time points prior and post RT. Images will be used to determine maps for functional lung avoidance and post-RT changes in the lung function and compared to standard-of-care assessment methods.

SUMMARY:
Cancer radiation treatment plans that employ lung functional avoidance methods require 3D maps that differentiate regions of healthy lung function from regions of compromised tissue to deliver sufficient dose to the tumor while preserving as much functioning lung as possible. Hyperpolarized xenon-129 MRI can provide maps of ventilatory function and gas exchange to the bloodstream. Improving treatment plans based on this novel imaging modality could reduce risk or severity of radiation pneumonitis and improve post-treatment quality of life.

DETAILED DESCRIPTION:
Customized 3D planning of radiation therapy for lung cancer delivers a lethal dose to the tumor region while avoiding important structures (spine) and organs (esophagus, heart, lungs). Since radiation dose to functioning lung is associated with acute radiation pneumonitis and chronic radiation fibrosis, researchers seek to shift dosage preferentially away from lung regions with highest function. Several lung functional imaging modalities have been investigated (ventilation-perfusion SPECT and PET, 4DCT, hyperpolarized 3He). These studies indicate that regional ventilation is not the optimal biomarker. What is needed is a high-resolution imaging modality, tolerable to patients who have difficulty holding their breath, that delineates regions of full lung function warranting preservation, and also identifies regions whose function is irrevocably gone.

The investigators propose a translational study applying Hyperpolarized Xenon (HXe) MRI to improve lung-health outcomes for lung cancer patients treated with radiation therapy. This study will focus on a patient cohort with significant heterogeneity: new patients with lung cancer and GOLD stage 3+ emphysema as a comorbidity and patients receiving RT for their second (primary) lung cancer. Optimizing radiation therapy treatment plans could provide a statistically significant benefit within a manageably small patient cohort. Maps will delineate three regions of functionality: regions of full function, having both ventilation and gas exchange to blood (where radiation should be reduced), regions where function is irrevocably absent (where radiation dose can be increased), and regions where function may be present or recoverable (where radiation should remain at the normal dose limit). In the first year the investigators will conduct an open-label Phase 1 clinical trial to optimize the hardware and functional imaging protocols, as well as generate and perform targeted RT treatment in a limited number of patients, with safety as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years with a diagnosis of non-small lung cancer and planned for a definitive course of radiation therapy.
* Preferred patients will have had successful radiation therapy for a prior lung cancer and developed a secondary lung cancer for which are to be treated.
* Other de-nuovo lung cancer patients planned for radiation therapy with lung heterogeneity from natural co-morbidities (e.g., COPD stage 3+).

Exclusion Criteria:

* Patients less than 18 years old
* Patients known to be pregnant - a positive pregnancy test will be used to respectively exclude pregnant patients,
* Any known contraindication to MRI examination
* Anyone with an implanted metal device
* Inability to provide informed consent
* A language, communication, cognitive or behavioral impairment that might interfere with fully informed participation in the study.
* History of uncompensated organ failure (i.e. organ failure that is not stabilized through medical intervention), which will be assessed by the PI.
* Homelessness or other unstable living situation
* Active drug or alcohol dependence
* Claustrophobia
* Subjects weighting more than 300 pounds.
* Subjects with chest size larger than the bore of MRI machine can accommodate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Number of patients reporting one or more adverse events related to hyperpolarized xenon inhalation in this population. | One year.
  Phase 1 will assess safety of inhaling hyperpolarized xenon in this patient population with severely affected lung function.

SECONDARY OUTCOMES:
Number of patients with radiation therapy related adverse events as assessed by CTCAE v4.0. | One year.
  First 10 patients enrolled in this study will have standard-of-care radiation therapy, and 10 more will have RT planned with functional lung avoidance maps based on HXe MRI. All patients will be monitored and followed for study related adverse events as assessed by CTCAE v4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States